CLINICAL TRIAL: NCT00790686
Title: Study of Tolerance and Effectiveness of Ureteral Stents MEMOKATH ® 051 in the Treatment of Chronic Strictures of the Ureter
Brief Title: Tolerance and Effectiveness of Ureteral Stents MEMOKATH ® 051 in Chronic Strictures of the Ureter
Acronym: TOTEME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2008/24
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Ureteral Obstruction
Keywords: Ureteral obstruction; Urologic surgical procedure; Stents; Endoscopy; Urology
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Memokath 051
  Interventions: Procedure: Insertion of Memokath 051

INTERVENTIONS:
Procedure: Insertion of Memokath 051 — Patients usually treated with double J stents will be included. The double J stent will be replaced by a MEMOKATH 051 stent under general anesthesia during a cystoscopy.

SUMMARY:
TOTEME offers to treat certain chronic strictures of the ureter with MEMOKATH 051 to assess its effectiveness, tolerance and mean durability during a 3 years follow up period.

Patients usually treated with double J stents will be included. The double J stent will be replaced by a MEMOKATH 051 stent under general anesthesia during a cystoscopy. After this procedure, the patients will have medical examinations, blood exams, radiography and renal sonography during 3 years. If a problem of tolerance or effectiveness is diagnosed, the ureteral stent MEMOKATH 051 will be changed or replaced with a double J stent.

DETAILED DESCRIPTION:
Introduction:

The chronic strictures of the ureter are usually treated by double J stents. They allow the emptying of the kidney and avoid the deterioration of renal function. Unfortunately, double J stents have to be replaced every 6 month and are at the origin of irritative lower urinary tract symptoms and lumbar pain which corrupt the quality of life of the patients.

Ureteral stricture could also be treated with MEMOKATH 051. These new ureteral stents seem not to require iterative changes and also not to cause irritative symptoms and lumbar pain. MEMOKATH 051 could therefore allow to reduce the number of changes and to ameliorate the quality of life of the patients.

Main objective:

Main objective is to assess effectiveness and tolerance of the MEMOKATH ® 051 in the treatment of chronic strictures of the ureter.

Resume:

Patients usually treated with double J stents will be included. The double J stent will be replaced by a MEMOKATH 051 stent under general anesthesia during a cystoscopy.

After this procedure, the patients will have medical examination, blood exams, radiography and renal sonography at 1 month, 3 month and every 6 month during a 3 years follow up period.

If a problem of tolerance or effectiveness is diagnosed, the ureteral stent MEMOKATH 051 will be changed or replaced with a double J stent and an adverse event will be declared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-year-old or superior
* Chronic stenosis of the ureter treated by placement of a ureteral endoprosthesis for more than six months;
* No possibility for surgical or endoscopic treatment of the ureteral stricture
* Free Consent, dated and signed by the patient
* Affiliated Subject of a regime of French national health and pensions organization.

Exclusion Criteria:

* Age under 18 year old
* Pregnant or nursing Women
* Patient having a life expectancy of less than 1 year
* Patient having unique kidney
* Patient having severe renal insufficiency (creatinin clearance under 30 ml/min)
* Possible surgical or endoscopic treatment of ureteral stricture
* Repeated urinary tract stones
* Urothelial tumor of the bladder
* Retro peritoneal fibrosis in the course of evolution
* Complications of double J stents requiring more thanks a lot every 6 months
* Against anaesthetic indication
* Lithiasic inlay probe Double J with obstruction within 6 months
* Persons put under maintenance of justice
* Persons in inability to understand the sequence of try

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Average durability of the stent MEMOKATH ® 051 | 3 years

SECONDARY OUTCOMES:
Proportion of ureteral stent MEMOKATH ® 051 positioning failure | 3 years
Average quality of life of the patients measured by auto-questionary | 3 years
Proportion of patients to which the ureteral stent was definitely taken away | 3 years
Expense of hospitalizations for replacement of the ureteral stent | 3 years
Proportion of replacement of the ureteral stent | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire Robert, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Department of Urology, University Hospital, Bordeaux, Bordeaux
  - Department of Urology, University Hospital, Limoges, Limoges
  - Department of Urology, Hospices Civils de Lyon, Lyon
  - Department of Urology, University Hospital, Toulouse, Toulouse

REFERENCES:
- [Background] Kulkarni R, Bellamy E. Nickel-titanium shape memory alloy Memokath 051 ureteral stent for managing long-term ureteral obstruction: 4-year experience. J Urol. 2001 Nov;166(5):1750-4. PMID 11586216
- [Background] Klarskov P, Nordling J, Nielsen JB. Experience with Memokath 051 ureteral stent. Scand J Urol Nephrol. 2005;39(2):169-72. doi: 10.1080/00365590510007720. PMID 16019773
- [Background] Pariente JL, Conort P. [Biomaterials used in contact with the urinary tract for urine drainage: catheters and ureteric stents]. Prog Urol. 2005 Nov;15(5):897-906. No abstract available. French. PMID 16475655
- [Background] Ringel A, Richter S, Shalev M, Nissenkorn I. Late complications of ureteral stents. Eur Urol. 2000 Jul;38(1):41-4. doi: 10.1159/000020250. PMID 10859440
- [Background] Kehinde EO, Rotimi VO, Al-Awadi KA, Abdul-Halim H, Boland F, Al-Hunayan A, Pazhoor A. Factors predisposing to urinary tract infection after J ureteral stent insertion. J Urol. 2002 Mar;167(3):1334-7. PMID 11832726
- [Background] Al-Kandari AM, Al-Shaiji TF, Shaaban H, Ibrahim HM, Elshebiny YH, Shokeir AA. Effects of proximal and distal ends of double-J ureteral stent position on postprocedural symptoms and quality of life: a randomized clinical trial. J Endourol. 2007 Jul;21(7):698-702. doi: 10.1089/end.2007.9949. PMID 17705753
- [Background] Hubner WA, Plas EG, Stoller ML. The double-J ureteral stent: in vivo and in vitro flow studies. J Urol. 1992 Aug;148(2 Pt 1):278-80. doi: 10.1016/s0022-5347(17)36572-2. PMID 1635117
- [Background] Poulsen AL, Schou J, Ovesen H, Nordling J. Memokath: a second generation of intraprostatic spirals. Br J Urol. 1993 Sep;72(3):331-4. doi: 10.1111/j.1464-410x.1993.tb00728.x. PMID 7693295
- [Background] Laaksovirta S, Valimaa T, Isotalo T, Tormala P, Talja M, Tammela TL. Encrustation and strength retention properties of the self-expandable, biodegradable, self-reinforced L-lactide-glycolic acid co-polymer 80:20 spiral urethral stent in vitro. J Urol. 2003 Aug;170(2 Pt 1):468-71. doi: 10.1097/01.ju.0000076389.88489.af. PMID 12853801
- [Background] Vaidyanathan S, Soni BM, Oo T, Sett P, Hughes PL, Singh G. Long-term result of Memokath urethral sphincter stent in spinal cord injury patients. BMC Urol. 2002 Nov 11;2:12. doi: 10.1186/1471-2490-2-12. Epub 2002 Nov 11. PMID 12427256
- [Background] Perry MJ, Roodhouse AJ, Gidlow AB, Spicer TG, Ellis BW. Thermo-expandable intraprostatic stents in bladder outlet obstruction: an 8-year study. BJU Int. 2002 Aug;90(3):216-23. doi: 10.1046/j.1464-410x.2002.02888.x. PMID 12133055
- [Background] Arya M, Mostafid H, Patel HR, Kellett MJ, Philp T. The self-expanding metallic ureteric stent in the long-term management of benign ureteric strictures. BJU Int. 2001 Sep;88(4):339-42. doi: 10.1046/j.1464-410x.2001.02322.x. PMID 11564017